CLINICAL TRIAL: NCT06832397
Title: Prospective Observational Study On the Detection of Peritoneal Metastases by Diagnostic LAparoscopy in Specific Subgroups of Patients With Locally Advanced Cervical canceR
Brief Title: Detection of Peritoneal Metastases by Diagnostic LAparoscopy in Patients With Locally Advanced Cervical Carcinoma
Acronym: SOLAR
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7386
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; Minimally invasive surgery in cervical cancer; Peritoneal metastases
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LACC patients with high-risk of peritoneal metastasis: Locally advanced cervical cancer patients with high-risk of peritoneal metastasis (AJCC stage T3/T4; grade 3 cervical cancer. all histotypes; FIGO stage IIIC2).
  Interventions: Procedure: Diagnostic laparoscopy

INTERVENTIONS:
Procedure: Diagnostic laparoscopy — Diagnostic laparoscopy with peritoneal biopsies

SUMMARY:
The study hypothesizes that specific subgroups of LACC patients, (AJCC stage T3/T4, grade 3 tumors, and para-aortic lymph node involvement), have a higher prevalence of peritoneal metastasis. This peritoneal spread may serve as a prognostic factor, and diagnostic laparoscopy could improve staging accuracy, thereby guiding personalized treatment strategies and improving oncological outcomes.

DETAILED DESCRIPTION:
Cervical cancer is the most prevalent gynecologic malignancy worldwide, with poor prognosis particularly in patients diagnosed with locally advanced cervical cancer (LACC; FIGO stage IB3-IVA). Although peritoneal metastasis is not included in FIGO staging, it is considered as a distant metastasis. Several studies have reported peritoneal disease in about 20% of LACC patients undergoing diagnostic laparoscopy, suggesting a potential role for laparoscopy in staging. However, the benefit of laparoscopy in surgical staging is controversial and the impact of peritoneal involvement on prognosis remains unclear.

This is a prospective, observational, single-center study. The primary objective is to assess the prevalence of peritoneal metastasis in specific subgroups of LACC patients (AJCC stage T3/T4, grade 3 cervical cancer, FIGO stage IIIC2) using diagnostic laparoscopy. Secondary objectives include evaluating 3-year disease-free survival (DFS), overall survival (OS), and treatment response rates to exclusive chemoradiotherapy (if pelvic peritoneal involvement, FIGO IVA) and chemo-immunotherapy (if upper abdominal peritoneal involvement, FIGO IVB) in patients with peritoneal metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Cervical cancer AJCC stage T3/T4 and/or
* Cervical cancer FIGO stage IB3 and IIA2-IVA grade 3 and/or
* Cervical cancer FIGO stage IIIC2 (para-aortic lymph node metastasis). Lymph node will be considered pathologic when the short axis diameter is > 10 mm at MRI scan and/or SUV max >2.5 at PET/CT-scan.
* All cervical histology sub-types will be included
* Stage assessment according to local Multidisciplinary Board
* Age >18 years
* Signature informed consent or substitute declaration on the consent form where applicable.

Exclusion Criteria:

* Patients with previous diagnosis of other cancers
* Performance status ECOG >2
* Pregnant women
* Contraindications to diagnostic laparoscopy
* Recurrent cervical cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients meeting the inclusion criteria
Study Population: Patients with newly diagnosed locally advanced cervical cancer at high risk of peritoneal metastases.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of peritoneal metastasis | 36 months after treatment
  Prevalence of peritoneal metastasis assessed by diagnostic laparoscopy

SECONDARY OUTCOMES:
3y-DFS | 36 months after treatment
  3 years disease free-survival
3y-OS | 36 months after treatment
  3 years overall survival
Response rate to CT-RT | 36 months after treatment
  Response rate to exclusive chemo-radiotherapy if IVA FIGO stage disease (only pelvic peritoneal disease, assessed by histological examination)
Response rate to CHT | 36 months after treatment
  Response rate to chemo-immunotherapy if IVB FIGO stage disease (upper abdomen peritoneal disease, assessed by histological examination)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolò Bizzarri, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome; Giovanni Scambia, Prof., Study Chair — Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome; Gabriella Ferrandina, Prof., Study Chair — Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome; Matteo Bruno, MD, Study Chair — Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome; Matteo Pavone, MD, Study Chair — Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome; Davide Arrigo, MD, Study Chair — Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
Locations (1):
- Policlinico Agostino Gemelli IRCCS, Rome, Italy

REFERENCES:
- [Background] Bizzarri N, Pedone Anchora L, Teodorico E, Certelli C, Galati G, Carbone V, Gallotta V, Naldini A, Costantini B, Querleu D, Fanfani F, Fagotti A, Scambia G, Ferrandina G. The role of diagnostic laparoscopy in locally advanced cervical cancer staging. Eur J Surg Oncol. 2024 Dec;50(12):108645. doi: 10.1016/j.ejso.2024.108645. Epub 2024 Aug 26. PMID 39214031
- [Background] de Foucher T, Bendifallah S, Ouldamer L, Bricou A, Lavoue V, Varinot J, Canlorbe G, Carcopino X, Raimond E, Monnier L, Graesslin O, Touboul C, Collinet P, Neveu ME, Huchon C, Darai E, Ballester M; Groupe de Recherche Francogyn, France. Patterns of recurrence and prognosis in locally advanced FIGO stage IB2 to IIB cervical cancer: Retrospective multicentre study from the FRANCOGYN group. Eur J Surg Oncol. 2019 Apr;45(4):659-665. doi: 10.1016/j.ejso.2018.11.014. Epub 2018 Dec 30. PMID 30685326
- [Background] Marnitz S, Kohler C, Roth C, Fuller J, Hinkelbein W, Schneider A. Is there a benefit of pretreatment laparoscopic transperitoneal surgical staging in patients with advanced cervical cancer? Gynecol Oncol. 2005 Dec;99(3):536-44. doi: 10.1016/j.ygyno.2005.07.005. Epub 2005 Aug 29. PMID 16126259
- [Background] Tewari KS, Sill MW, Penson RT, Huang H, Ramondetta LM, Landrum LM, Oaknin A, Reid TJ, Leitao MM, Michael HE, DiSaia PJ, Copeland LJ, Creasman WT, Stehman FB, Brady MF, Burger RA, Thigpen JT, Birrer MJ, Waggoner SE, Moore DH, Look KY, Koh WJ, Monk BJ. Bevacizumab for advanced cervical cancer: final overall survival and adverse event analysis of a randomised, controlled, open-label, phase 3 trial (Gynecologic Oncology Group 240). Lancet. 2017 Oct 7;390(10103):1654-1663. doi: 10.1016/S0140-6736(17)31607-0. Epub 2017 Jul 27. PMID 28756902
- [Background] Monk BJ, Colombo N, Tewari KS, Dubot C, Caceres MV, Hasegawa K, Shapira-Frommer R, Salman P, Yanez E, Gumus M, Olivera Hurtado de Mendoza M, Samouelian V, Castonguay V, Arkhipov A, Tekin C, Li K, Keefe SM, Lorusso D; KEYNOTE-826 Investigators. First-Line Pembrolizumab + Chemotherapy Versus Placebo + Chemotherapy for Persistent, Recurrent, or Metastatic Cervical Cancer: Final Overall Survival Results of KEYNOTE-826. J Clin Oncol. 2023 Dec 20;41(36):5505-5511. doi: 10.1200/JCO.23.00914. Epub 2023 Nov 1. PMID 37910822